CLINICAL TRIAL: NCT03994926
Title: Evaluation of an Eye Tracking Sensor to Detect Cannabis Impairment
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID-19 Pandmic halted study
Sponsor: Battelle Memorial Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 131310
Record Dates: First submitted 2019-06-12; First posted 2019-06-21 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cannabis Intoxication
Keywords: cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Directed smoking of about 3.6% THC cannabis cigarette
  Interventions: Device: Virtual Reality Eye Tracking after smoking Cannabis - HTC Vive Pro-Eye; Drug: Cannabis cigarette - 4.0% THC

INTERVENTIONS:
Device: Virtual Reality Eye Tracking after smoking Cannabis - HTC Vive Pro-Eye — Device measures smooth eye pursuit and response to light flash after pt smokes cannabis
Drug: Cannabis cigarette - 4.0% THC — smoked cannabis 4.0% THC
  Other Names: Marijuana

SUMMARY:
The purpose of this study is to determine if an eye tracking impairment sensor can detect cannabis-induced impairment after using cannabis.The overall objective is to correlate measures collected from the eye tracking sensor with measures related to cannabis impairment (e.g., plasma THC levels, self-reported cannabis subjective effects, cognitive effects).

DETAILED DESCRIPTION:
The proposed project is a single-visit clinical laboratory study to evaluate the initial efficacy of an eye tracking sensor to detect cannabis-related impairment.

Participants will be experienced but not frequent cannabis users without evidence of heavy alcohol or illicit drug use or other physical or mental health illness. Participants will come in for one screening visit, and those who consent, are eligible, and enroll will complete one experimental laboratory session involving smoking of 50% of 1 active (approximately 4.0% THC) cannabis cigarette. Assessments will be collected after-cannabis smoking up to 4 hours. Participants will be sent home from the laboratory via taxi.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign a confidentiality agreement stating the will not discuss study specifics, information or materials presented to them in the study with those not involved in the study;
2. Currently living in Baltimore City or Baltimore County, MD, or Investigator discretion;
3. Able to read, understand, and sign informed consent;
4. 18-55 years old;
5. Self-reports lifetime smoking of cannabis at least 10 times without any negative side effects;
6. Self-reports past-year smoking of cannabis at least 1 time but no more than 2 days per week on average;
7. Designation of Medically Healthy for Research by the Study Physician.
8. Agree to abstain from consuming alcohol for 10 hours and marijuana for 72 hour prior to the study visit

Exclusion Criteria:

1. BAC > 0.020% as measured by alcohol breathalyzer;
2. Meets DSM-5 criteria for any current Axis I disorder other than mild or moderate Cannabis Use Disorder;
3. Self-reported current desire to stop cannabis use, defined as 7 or greater on an 11-rung (scale of 0-10) on the Contemplation Ladder assessment;
4. Self-reported current asthma, chronic obstructive pulmonary disease, hypertension, cardiovascular disease or any other medical illness that precludes participation based on the clinical judgment of the Study Physician and Investigative Team;
5. Has difficulties with blood draws or poor venous access;
6. History of blood donation in the past 30 days or receiving blood products within the past 2 months prior to any experimental visit;
7. Investigator discretion due to self-reported use of medical cannabis or using cannabis for self-medication;
8. Among females, current pregnancy or lactation or attempting to get pregnant, or at risk of becoming pregnant, as defined as being sexually active with a male partner and not willing to use a reliable form of contraception;
9. Investigator discretion due to use of caffeine, over-the-counter (OTC) drugs, prescription drugs, alcohol, or physical/mental health history;
10. Positive urine drug screen for drugs included on the urine drug panel other than cannabis;
11. Acute illness (such as cold or flu) which will require participant to be rescheduled, if authorized by study PI;
12. Vital signs thought to be clinically significant by licensed medical professional;
13. Self-reported history or medical evidence of prior intravenous drug use; and
14. Investigator discretion due to medical, mental health, or substance use history.
15. Presence of implanted devices in the body (pacemaker etc)
16. Previously reported negative effects from the use of VR goggles or negative effects from the use of VR goggles during screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pupil Dilation | Before and after smoking (up to 240 minutes)
  Change in pupil dilation in different lights will be measured by the eye tracking sensor
Change from baseline in Gaze Nystagmus | Before and after smoking (up to 240 minutes)
  Change in Gaze Nystagmus will be measured by the eye tracking sensor
Change from baseline in Lack of Convergence | Before and after smoking (up to 240 minutes)
  Change in Lack of Convergence will be measured by the eye tracking sensor

SECONDARY OUTCOMES:
Plasma THC | Before and after smoking (9 timepoints up to 240 minutes post smoking)
  Plasma concentration before and after smoking
Change from baseline in Cannabis Subjective Effects | Before and after smoking (up to 240 minutes post smoking)
  Scores for the question "do you feel a drug effect" are measured on a 0-100 point visual analogue scale to measure change in marijuana intoxication across timepoints.
Change from baseline in Four Choice Reaction Time Task | Before and after smoking (up to 240 minutes post smoking)
  Will assess changes in psychomotor/cognitive performance known to be sensitive to the acute effects of smoked cannabis.
Change from baseline in Digit Symbol Substitution Task | Before and after smoking (up to 240 minutes post smoking)
  Will assess changes in psychomotor/cognitive performance known to be sensitive to the acute effects of smoked cannabis.

CONTACTS AND LOCATIONS:
Locations (1):
- Battelle Memorial Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casswell S, Marks D. Cannabis induced impairment of performance of a divided attention task. Nature. 1973 Jan 5;241(5384):60-1. doi: 10.1038/241060b0. No abstract available. PMID 4696937
- [Background] Desrosiers NA, Ramaekers JG, Chauchard E, Gorelick DA, Huestis MA. Smoked cannabis' psychomotor and neurocognitive effects in occasional and frequent smokers. J Anal Toxicol. 2015 May;39(4):251-61. doi: 10.1093/jat/bkv012. Epub 2015 Mar 4. PMID 25745105
- [Background] Murillo R, Crucilla C, Schmittner J, Hotchkiss E, Pickworth WB. Pupillometry in the detection of concomitant drug use in opioid-maintained patients. Methods Find Exp Clin Pharmacol. 2004 May;26(4):271-5. PMID 15319805
- [Background] Pickworth WB, Rohrer MS, Fant RV. Effects of abused drugs on psychomotor performance. Exp Clin Psychopharmacol. 1997 Aug;5(3):235-41. doi: 10.1037//1064-1297.5.3.235. PMID 9260070